CLINICAL TRIAL: NCT07020208
Title: Novice Nurses Preparation for Clinical Practice: Examining the Impact of Transition Shock Readiness Skills on Career Entrenchment, and Interprofessional Readiness
Brief Title: Ovice Nurse Transition Shock and Readiness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Port Said University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 111-h
Record Dates: First submitted 2025-05-28; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Nurses
Keywords: Novice Nurses Newly Graduated Nurses Transition to Practice Transition Shock Clinical Practice Readiness

STUDY DESIGN:
Intervention Model Description: open-label, two-arm Randomized Control Trail (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nterventional study (Experimental): Description: the participated nurses will receive session about Transition Shock Readiness skills
  Interventions: Behavioral: Transition Shock skills
- control group (No Intervention)

INTERVENTIONS:
Behavioral: Transition Shock skills — * Assign experienced nurse mentors to new graduates.
  * Conduct weekly one-on-one meetings for the first three months, then biweekly for ongoing support.
  * Discuss challenges, successes, and strategies for coping with difficult situations.
  * Provide case study reviews where mentors guide mentees through real-world nursing scenarios.
    * Skills Applied: interpersonal communication. 2. Peer Support Groups
    * Content:
  * Establish weekly or biweekly group discussions where nurses share challenges and coping strategies.
  * Use reflective journaling prompts to encourage discussion.
  * Introduce role-playing exercises for dealing with complex patients, staff conflicts, and ethical dilemmas.
  Arms: nterventional study

SUMMARY:
This study aims to investigate the impact of a transition shock program on career entrenchment and readiness for interprofessional learning among newly graduated nurses.

DETAILED DESCRIPTION:
This study aims to investigate the impact of a transition shock program on career entrenchment and readiness for interprofessional learning among newly graduated nurses.

Hypotheses:

H1: After the intervention, the study group will report significantly lower transition shock scores compared to the control group.

H2: After the intervention, the study group will report significantly lower career entrenchment scores compared to the control group.

H3: After the intervention, the study group will report significantly higher readiness for interprofessional learning scores compared to the control group.

H4: There will be a significant interaction effect between time (pre-test vs. post-test) and group (study vs. control), where the study group will show greater improvement in readiness for interprofessional learning and greater reduction in transition shock and career entrenchment compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* 1. Newly employed nurses who have worked for less than six months in the profession.

  2. Nurses who have not received prior transition-related training before participation in the study.

  3. Nurses willing to participate voluntarily and provide informed consent.

Exclusion Criteria:

1. Nurses with previous work experience before their current job.
2. Those who decline participation or withdraw from the study.
3. Nurses enrolled in ongoing professional development programs related to transition or interprofessional education.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-02 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Transition Shock Readiness skills of nurses | 3 monthes
  Change From Baseline in Transition Shock Readiness Score at the end of the intervention period

IPD SHARING:
Plan to Share IPD: Yes